CLINICAL TRIAL: NCT02442245
Title: The Effect of XSurgeTM Supplementation on Biomarkers, Oxidative Stress, and Recovery From High Intensity Resistance Exercise
Brief Title: The Effect of XSurge Supplementation on Biomarkers and Performance From High Intensity Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kemin Foods LC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 14HUS002
Record Dates: First submitted 2015-04-30; First posted 2015-05-13 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Exercise Performance Recovery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Placebo group will receive microcrystalline cellulose
  Interventions: Other: Placebo: Microcrystalline Cellulose
- Treatment (Active Comparator): Treatment group will get 2 g daily of XSurge in microcrystalline cellulose
  Interventions: Dietary Supplement: XSurge
- Control Group (Sham Comparator): The control group will be included to quantify or describe the effects of the acute exercise training but will not receive any supplement
  Interventions: Other: Control: No supplementation

INTERVENTIONS:
Dietary Supplement: XSurge — During part one of the study, 28 days of supplementation with XSurge will be provided. During the second part of the study 6 weeks of supplementation with XSurge will accompany a training program.
  Arms: Treatment
Other: Placebo: Microcrystalline Cellulose
  Arms: Placebo
Other: Control: No supplementation
  Arms: Control Group

SUMMARY:
Part one of this study will consist of baseline (BL) testing, 28 days of daily supplementation with XSurge, and an exercise protocol. The acute exercise protocol consists of five visits, of which, the first visit will consist of maximal strength testing. The remaining visits will consist of performance testing and muscle evaluation.

Phase two of this study will consist of six weeks of supervised resistance training along with supplementation of XSurge. Following the six weeks of training, subjects will complete a second acute exercise protocol. Measures to be evaluated will consist of performance testing and muscle evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active.
* Subject is judged by the Investigator to be healthy and free of any physical limitations
* Subject is male 18-35 y of age, inclusive
* Subject has a body mass index of 18.0-34.9 kg/m2
* Subject is willing to maintain habitual diet
* Subject is willing to abstain from dietary supplementation
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators

Exclusion Criteria:

* Subject is currently or will be enrolled in another clinical trial.
* Subject has a history or presence of a clinically relevant cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorder.
* Subject has a history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Subject is unable to perform physical exercise
* Subject is a current smoker or has quit within the last 6 months
* Subject is engaged in an extreme diet including but not limited to, Atkins, South Beach, Intermittent Fasting, etc.
* Subject is allergic to the study product or placebo
* Subject is taking any other nutritional supplement or performance enhancing drug
* Subjects that have donated blood or plasma within the previous week
* Subject has any chronic illness that causes continuous medical care
* Taking any type of prescription or over-the-counter medication including but not limited to corticosteroids, non-steroidal anti-inflammatory drugs, and antibiotics within the 14 days prior to the screening visit.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Strength as measured by Peak Torque (Biodex) | Part 1-Change from baseline after 28 days of supplementation; Part 2-Change from baseline after 6 weeks of supplementation plus exercise
Biomarkers (Cortisol and Creatine Phosphokinase) | Part 1-Change from baseline after 28 days of supplementation; Part 2-Change from baseline after 6 weeks of supplementation plus exercise

SECONDARY OUTCOMES:
Subjective Feelings of Recovery (Likert Scale) | Part 1-Change from baseline after 28 days of supplementation; Part 2-Change from baseline after 6 weeks of supplementation plus exercise
Muscle Soreness (VAS) | Part 1-Change from baseline after 28 days of supplementation; Part 2-Change from baseline after 6 weeks of supplementation plus exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

REFERENCES:
- [Derived] Jajtner AR, Townsend JR, Beyer KS, Varanoske AN, Church DD, Oliveira LP, Herrlinger KA, Radom-Aizik S, Fukuda DH, Stout JR, Hoffman JR. Resistance Exercise Selectively Mobilizes Monocyte Subsets: Role of Polyphenols. Med Sci Sports Exerc. 2018 Nov;50(11):2231-2241. doi: 10.1249/MSS.0000000000001703. PMID 29957728